CLINICAL TRIAL: NCT02229695
Title: The Effect of Different Types of Temporary Abdominal Closure on Intra Abdominal Hypertension and Abdominal Compartment Syndrome.
Brief Title: The Effect of Different Types of Temporary Abdominal Closure on Intra Abdominal Hypertension.
Acronym: TACACS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Gad Shaked MD, Professor, Soroka University Medical Center
Other Study IDs: SOR-0167-14
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Intra Abdominal Hypertension; Abdominal Compartment Syndrome
Keywords: Trauma; Sepsis; Temporary abdominal closure; Bogota bag; Vacuum assisted closure
MeSH Terms: conditions — Intra-Abdominal Hypertension; Wounds and Injuries; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective comparison trial. Patients that will be included in the trial are those that will have operations in which their abdominal closure is temporary, i.e. patients sustaining trauma or septic abdomen.

Patients will be grouped according to the method of temporarily abdominal closure (TAC) procedure:

1. Vacuum-assisted closure (VAC)
2. "Bogota bag" (BB), a sterile intravenous bag silo closure. The two methods are currently accepted with no clear cut evidence to prefer one on another. At Soroka Medical Center the decision to choose either of the methods is at the surgeon's discretion.

Intra-abdominal pressure will be measured in all patients by the urinary bladder pressure technique at 6 12 24 ant 48 hours post operation. The measurement is a routine procedure done as part of the monitoring processes of critically ill patients in the General Intensive Care Unit (GICU).

Patients will be evaluated for the development of acute intra abdominal hypertension with or without abdominal compartment syndrome.

DETAILED DESCRIPTION:
Comparison of intra-Abdominal hypertension development after bogota bag or VAC abdominal closure Protocol

Trial objective:

To investigate and compare in a standardized manner the development of intra-abdominal hypertension (IAH) following VAC closure and "Bogota bag".

Study design:

This is a prospective comparison trial. Patients that will be included in the trial are those that will have operations in which their abdominal closure is temporary, i.e. patients sustaining trauma or septic abdomen.

Patients will be grouped according to the method of temporarily abdominal closure (TAC) procedure:

1. VAC closure
2. "Bogota bag" (BB), a sterile intravenous bag silo closure. The two methods are currently accepted with no clear cut evidence to prefer one on another. At Soroka Medical Center the decision to choose either of the methods is at the surgeon's discretion.

Intra-abdominal pressure will be measured in all patients by the urinary bladder pressure technique at 6 12 24 ant 48 hours post operation. The measurement is a routine procedure done as part of the monitoring processes of critically ill patients in the GICU. It will be carried out by a nurse who will be blinded as to the type of the abdominal closure.

Patients will be evaluated for the development of acute and significant respiratory compromise, including an elevated inspiratory pressure of >35 mbar and a decreased partial oxygen pressure / fraction of inspired oxygen (PaO2/FIO2) of <150 torr, hypotension (<90 mmHg systolic pressure not due to hemorrhagic, septic, or neurogenic causes), renal dysfunction (urine output, <30 mL/hr), and a clinically determined rigid, tense abdomen, and increased abdominal circumference.

The following data will be recorded. Hemodynamics (mean arterial pressure, heart rate), lactate, PaO2, partial carbonic dioxide pressure (PaCO2), tidal volume, peak airway pressure) and renal (urine output) functions will be registered at 24 and 48 hours following surgery).

Data on the indication for operation, type of trauma, its severity and the operative procedures.

Acute Physiologic and Chronic Health Evaluation II (APACHE II) and fluid balance at 24 and 48 hours.

Reoperations. Time in ICU and time to final abdominal closure.

Study population:

All patients with severe abdominal trauma or none traumatic acute abdomen, that at the end of operation the surgeon will decide to use temporary abdominal closure (TAC).

Inclusion Criteria Adults male or female over 18 years old. The surgeon decides the need for TAC at the end of operation.

Exclusion Criteria Patients that the surgeon estimates they will not survive 24 hours.

End points:

Development of IAH Development of abdominal compartment syndrome (ACS) Need for reoperation of decompressive laparotomy during first 48 hours. Time to final (on discharge from hospital) abdominal closure and the type of closure.

Statistical methodology The calculated sample size based on power of 0.80, alpha 0.05, known incidence of 0.25 and estimated incidence of 0.10 is 42 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults male or female over 18 year old undergoing emergency laparotomy. Patients that have their abdominal wall closed at the end of surgery by a temporary closure technique.

Exclusion Criteria:

* Patients that according to the surgeon estimates will not survive 24 hours.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that undergo emergent laparotomy for trauma or non-traumatic surgical emergency condition, and that according to the surgeon decision get their abdominal wall closed by a temporary closure technique.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Intra abdominal hypertension | 48 hours
  measured via a Foley catheter

SECONDARY OUTCOMES:
Abdominal compartment syndrome | 48 hours
  According to clinical signs (hypotension, increased inspiratory pressure, decreased urinary output).

CONTACTS AND LOCATIONS:
Overall Officials: Gad Shaked, Prof., Principal Investigator — Soroka University Medical Center